CLINICAL TRIAL: NCT02622425
Title: The Effect of the Carotenoid-producing Bacillus Strain PD01 on Cardiovascular Health and Microbial Environment
Brief Title: The Effect of PD01 on Cardiovascular Health and Microbial Environment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bouke Salden, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 153001
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Overweight; Obesity
Keywords: Carotenoid; Bacillus; Microbiota; Cardiovascular health
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PD01 (Active Comparator): Carotenoid-producing Bacillus strain PD01
  Interventions: Dietary Supplement: PD01
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — maltodextrin
  Arms: Placebo
Dietary Supplement: PD01 — Carotenoid-producing Bacillus strain PD01
  Arms: PD01

SUMMARY:
This randomized, placebo-controlled trial aims to determine the effects of daily administration of a carotenoid-producing Bacillus strain PD01 over a 6-week period on cardiovascular health biomarkers, microbiota composition and functioning and intestinal barrier function in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men/women (BMI 25-35 kg/m2)
* Healthy individuals
* Age between 18 and 70 years
* Fasting glucose < 7.0 mmol/L
* Normal HbA1c (4.4 to 6.2%)

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L);
* History of (severe) cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
* Abdominal surgery interfering with gastrointestinal function, upon judgment of the principle investigator)
* Use of medication interfering with endpoints
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Use of antibiotics in the 90 days prior to the start of study
* Known pregnancy, lactation
* Abuse of products; alcohol (> 20 alcoholic consumptions per week) and drugs
* Smoking
* Blood donation within 3 months before study period
* Plans to lose weight or following a hypocaloric diet during the study period;
* Weight gain or loss > 3 kg in previous 3 months
* High physical activity (>4.5 hours of running/week)
* Hormone replacement therapy (women)
* History of any side effects towards intake of pro- or prebiotic supplements of any kind
* History of any side effects towards intake of carotenoids
* Prohibited use of pro-, pre- or synbiotics during study period and from one month prior to start of study.
* High intake of fruits and vegetables (more than the 75th percentile of dietary intake of fruits and vegetables)
* Vegetarians/vegans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect on lipid peroxidation measured urinary F2-isoprostane excretion | 6 weeks
  The primary objective of this study is to evaluate the efficacy of PD01 on lipid peroxidation by measuring F2-isoprostane excretion in 24-hour urine, after 6 weeks of administration.

SECONDARY OUTCOMES:
Effect on lipid peroxidation measured by blood concentration of F2-isoprostanes | 6 weeks
Effect on lipid peroxidation measured by blood total antioxidant capacity | 6 weeks
Effect on lipid peroxidation measured by blood MDA concentration | 6 weeks
Effect on low-grade inflammation measured by blood concentration of TNFalfa | 6 weeks
Effect on platelet aggregation measured by blood concentration of P-selectin | 6 weeks
Effect on blood glucose concentrations measured by blood glucose concentration | 6 weeks
Effect on blood lipid profile | 6 weeks
Effect on blood pressure | 6 weeks
Effect on body composition measured by BMI | 6 weeks
Effect on body composition measured by waist-hip circumference (WHC) | 6 weeks
The effect on fecal microbial community composition measured by fecal microbial community composition | 6 weeks
The effect on fecal microbial community composition measured by fecal short chain fatty acids (SCFA) | 6 weeks
Effect on gut barrier function measured by a sugar test | 6 weeks
To assess the bioavailability of PD01 by measuring blood carotenoid concentration | 6 weeks
Effect on digestive tolerance measured by GSRS questionnaire | 6 weeks
Effect on digestive tolerance measured by Bristol Stool Chart | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands